CLINICAL TRIAL: NCT01415947
Title: V-Chordal Adjustable System for Chordal Replacement in Mitral Valve Insufficiency Due to Leaflet Prolapse
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company business decision
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH1-1
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Mitral Leaflet Prolapse
Keywords: Heart disease; Device; Mitral valve; leaflet prolapse; Heart valve disease; Cardiovascular disease; Neochordae
MeSH Terms: conditions — Mitral Valve Prolapse; Heart Diseases; Heart Valve Diseases; Cardiovascular Diseases

INTERVENTIONS:
Device: V Chordal — V-Chordal system, consists in the ability to adjust (elongate or shorten) the neochordae "off-pump" . The adjustment mechanism allows overcoming the main problem of chordal replacement by enabling accurate sizing of the chords.

SUMMARY:
The V-Chordal System is a new technology for mitral repair. The Valtech V-Chordal system, consists in the ability to adjust (elongate or shorten) the neochordae "off-pump" to achieve an optimal coaptation. The adjustment mechanism allows overcoming the main problem of chordal replacement by enabling accurate sizing of the chords.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Degenerative mitral insufficiency with mitral leaflet prolapsed , who are candidates for mitral valve repair according to ESC or ACC/AHA guidelines.
* Patient able and willing to return to the implant center for follow-up visits
* Able and willing to give informed consent and follow protocol procedures.

Exclusion Criteria:

* Inadequate echocardiographic window for transthoracic imaging
* Severe organic lesions with retraction of chordate tendineae, severly fibrotic and immobile leaflets, severely deformed subvalvular apparatus.
* Evolving endocarditis or active endocarditis in the last 3 months.
* Heavily calcified annulus or leaflets.
* Congenital malformation with limited valvular tissue
* Patient requires mitral valve replacement.
* Previously implanted annuloplasty ring/band.
* Patient requires aortic or pulmonic valve replacement or repair.
* Patient is pregnant (urine HCG test result positive) or lactating.
* Patient has a major cardiac or non-cardiac disease, which in the investigator's experience produces an unacceptable surgical risk.
* Life expectancy of less than twelve months.
* Patient is participating in concomitant research studies of investigational products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Technical success rate | 6 months
  ability to:
  1. Anchor the system in the papillary muscle;
  2. Suture the leaflet;
  3. Release the V-Chordal system and extract the delivery system with no lesions to adjacent tissue.
  4. Technical feasibility of chordal length adjustment. When required, adjustment of chords after weaning from CPB
Efficacy | 30 days and 6 months
  The ability of the V-Chordal System to correct leaflet prolapse of the treated segments as assessed by echordiography. Correction is defined as leaflet displacement <2 mm above the annulus in the septolateral view.

SECONDARY OUTCOMES:
Incidence of Major Adverse Events (MAE). | 30 days, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ottavio Alfiieri, MD, Principal Investigator — Hospital San Raffaele
Locations (1):
- HSR, Milan, Italy